CLINICAL TRIAL: NCT00888888
Title: Risk Factors for Colonic Resections in Patients With Suspected Acute Appendicitis
Brief Title: Colonic Resections in Patients With Suspected Appendicitis
Status: Completed | Type: Observational
Sponsor: Cirujanos la Serena (Other)
Responsible Party: Principal Investigator, MARCELO A. BELTRAN, M.D., DIGESTIVE SURGEON, Cirujanos la Serena
Other Study IDs: HLS-2604009-01
Record Dates: First submitted 2009-04-27; First posted 2009-04-28 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Colectomy; Appendicitis
Keywords: Acute appendicitis; Colonic diverticulitis; Colonic tumors; Colonic resections
MeSH Terms: conditions — Appendicitis; Diverticulitis, Colonic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort: Patients with colonic resections: Colonic resections in patients submitted to appendicectomy for suspected acute appendicitis
  Interventions: Procedure: Right hemicolectomy with or without primary anastomosis

INTERVENTIONS:
Procedure: Right hemicolectomy with or without primary anastomosis — During open classic appendectomy (McBurney incision) the surgeon decided to convert to midline extended laparotomy to perform a right hemicolectomy

SUMMARY:
Although many reports have been published on colonic resections in patients with suspected appendicitis and the diseases that cause the decision to resect the colon have been identified and their proper treatments have been established, there is no report on the risk factors present in converting a simple appendectomy into a major colonic resection.

The investigators aimed to identify the risk factors that lead the surgeon to perform a colonic resection in patients undergoing surgery for initially suspected acute appendicitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 15 years of age
* Male or female
* Suspected of having acute appendicitis
* Converted to right hemicolectomy

Exclusion Criteria:

* Patients in whom a right hemicolectomy was planned initially
* Right hemicolectomy for causes other than suspected acute appendicitis

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients submitted to appendectomy for suspected acute appendicitis and in whom the surgeon takes the decision to convert to right colectomy based on operative findings and other factors the we aim to identify
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2009-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Short-term survival | 3 months

SECONDARY OUTCOMES:
Long-term survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: MARCELO A BELTRAN, M.D., Principal Investigator — Hospital de La Serena
Locations (1):
- Hospital de La Serena, La Serena, Coquimbo Region, Chile